CLINICAL TRIAL: NCT00069316
Title: A Phase I/II Randomized, Placebo-Controlled Trial to Assess the Safety and Efficacy of Intravenous Immunoglobulin G (Omr-IgG-am) Containing High Anti-West Nile Virus Antibody Titers in Patients With, or at High Risk for Progression to West Nile Virus(WNV)
Brief Title: Omr-IgG-am(Trademark) for Treating Patients With or at High Risk for West Nile Virus Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: NIAID, DMID
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 030306; 03-CC-0306
Record Dates: First submitted 2003-09-22; First posted 2003-09-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-02-18

CONDITIONS: West Nile Virus
Keywords: West Nile Virus; Encephalitis; Virus; Mosquito; Fever; WNV; Myelitis
MeSH Terms: conditions — Encephalitis; Virus Diseases; Fever; Myelitis

INTERVENTIONS:
Drug: Omr-IgG-am

SUMMARY:
Investigators will assess whether Omr-IgG-am(Trademark), an intravenous immunoglobulin (IVIg) containing antibodies specific for West Nile virus (WNV), is safe and well-tolerated in patients with suspected or laboratory diagnosed WNV disease. An initial estimation of efficacy will also be made.

This Phase I/II study will enroll hospitalized adults with a presumptive diagnosis of West Nile encephalitis and/or myelitis or those with a positive laboratory test for diagnosis of WNV infection who are at high risk for progressing to severe neurologic disease based on age or immunosuppression. Patients will be randomized in blocks of five to receive either Omr-IgG-am(Trademark), Polygam(Registered Trademark) S/D (IVIG containing minimal anti-WNV antibodies) or normal saline in a ratio of 3:1:1. Patients and investigators will be blinded to treatment assignments.

Patients will receive a single intravenous dose of study medication or one of two placebos. The study participants will receive 0.5 grams/kg of Omr-IgG-am(Trademark) or Polygam(Registered Trademark) S/D or a comparable volume of normal saline. All patients will be followed for safety, natural history endpoints, and efficacy. A subset of patients will have pharmacokinetic measurements of specific anti- WNV antibodies assessed following treatment.

The primary endpoints are safety and tolerability following Omr-IgG-am(Trademark) administration.

Secondary endpoints include pharmacokinetics of specific anti-WNV antibodies, mortality in confirmed WNV positive patients, and the combination of mortality and functional status at three months in both confirmed WNV-infected patients and all patients by intention to treat. This combined endpoint will be measured using four standardized measures of cognitive and functional status: the Barthel Index; the Modified Rankin Scale; the Glasgow Outcome Score; and the Modified Mini-Mental Status Examination. A comparison of outcomes will be made for the group receiving Omr-IgG-am(Trademark) versus those receiving either placebo, and between the two placebo groups. Other secondary endpoints include the proportion of patients in each group returning to pre-morbid baseline and each subject's improvement at 3 months as compared to that subject's worst (of any previous) evaluation.

Natural history endpoints will also be assessed. They will include the duration of intensive care unit (ICU) and hospital stay, development and persistence of WNV-specific IgG and IgM antibodies, combined functional score and mortality at 3 months between the group with encephalitis and/or myelitis at baseline versus the group with a positive WNV test only, outcomes in patients treated late in coma and correlation of outcome with time-to-treatment following symptom onset.

DETAILED DESCRIPTION:
Investigators will assess whether Omr-IgG-am(Trademark), an intravenous immunoglobulin (IVIg) containing antibodies specific for West Nile virus (WNV), is safe and well-tolerated in patients with suspected or laboratory diagnosed WNV disease. An initial estimation of efficacy will also be made.

This Phase I/II study will enroll hospitalized adults with a presumptive diagnosis of West Nile encephalitis and/or myelitis or those with a positive laboratory test for diagnosis of WNV infection who are at high risk for progressing to severe neurologic disease based on age or immunosuppression. Patients will be randomized in blocks of five to receive either Omr-IgG-am(Trademark), Polygam(Registered Trademark) S/D (IVIG containing minimal anti-WNV antibodies) or normal saline in a ratio of 3:1:1. Patients and investigators will be blinded to treatment assignments.

Patients will receive a single intravenous dose of study medication or one of two placebos. The study participants will receive 0.5 grams/kg of Omr-IgG-am(Trademark) or Polygam(Registered Trademark) S/D or a comparable volume of normal saline. All patients will be followed for safety, natural history endpoints, and efficacy. A subset of patients will have pharmacokinetic measurements of specific anti- WNV antibodies assessed following treatment.

The primary endpoints are safety and tolerability following Omr-IgG-am(Trademark) administration.

Secondary endpoints include pharmacokinetics of specific anti-WNV antibodies, mortality in confirmed WNV positive patients, and the combination of mortality and functional status at three months in both confirmed WNV-infected patients and all patients by intention to treat. This combined endpoint will be measured using four standardized measures of cognitive and functional status: the Barthel Index; the Modified Rankin Scale; the Glasgow Outcome Score; and the Modified Mini-Mental Status Examination. A comparison of outcomes will be made for the group receiving Omr-IgG-am(Trademark) versus those receiving either placebo, and between the two placebo groups. Other secondary endpoints include the proportion of patients in each group returning to pre-morbid baseline and each subject's improvement at 3 months as compared to that subject's worst (of any previous) evaluation.

Natural history endpoints will also be assessed. They will include the duration of intensive care unit (ICU) and hospital stay, development and persistence of WNV-specific IgG and IgM antibodies, combined functional score and mortality at 3 months between the group with encephalitis and/or myelitis at baseline versus the group with a positive WNV test only, outcomes in patients treated late in coma and correlation of outcome with time-to-treatment following symptom onset.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to participate in this clinical trial, all subjects (or legal representative) must provide written informed consent. Only patients meeting entry criteria will be enrolled. Eligible subjects must fall into one of two categories:

A. Hospitalized patients greater than or equal to 18 years of age with encephalitis and/or myelitis as defined below:

New neurologic abnormality:

Asymmetric extremity weakness without sensory abnormality; or

Other neurologic abnormality (including altered level of consciousness, dysarthria and dysphagia) plus fever (subjective or objective) within the previous 4 days

AND

CSF examination within the previous 96 hours showing:

Absence of organism on gram or fungal stain

White blood cell count greater than or equal to 4 per mm(3) corrected for significant red blood cell contamination.

Ratio of CSF: plasma glucose of greater than or equal to 40% (CSF glucose/plasma glucose greater than or equal to 0.4)

OR

B. Hospitalized patients without encephalitis and/or myelitis as defined below who meet the following criteria:

A positive IgM serology or PCR test for WNV in blood or cerebrospinal fluid,

AND

Clinical illness compatible with WNV infection as described by occurrence of greater than or equal to 3 of the following findings during the preceding less than or equal to 10 days:

Diarrhea, headache, fever greater than 38 degrees Celsius, nausea and/or vomiting, myalgias and/or arthralgias, nuchal rigidity, macular or papular rash, new neurological abnormality

AND

A risk factor for the development of WNV neurologic disease as defined by:

Age greater than or equal to 40 years, or

Age greater than or equal to 18 years, plus immunosuppression, as defined by any of the following:

Hematologic malignancy, previous diagnosis of diabetes mellitus, chemotherapy within previous 4 weeks, stem cell transplant recipient or solid organ transplant recipient, taking immunosuppressive medications, including prednisone greater than or equal to 7.5 mg/day within the previous 4 weeks, history of human immunodeficiency virus (HIV) infection, congenital immunodeficiency syndrome (including common variable immunodeficiency)

EXCLUSION CRITERIA:

Unable to obtain valid informed consent

History of intolerance (including anaphylaxis) to IVIg or related compounds

Known history of IgA deficiency

Known history of hypersensitivity to maltose.

History of (or at time of study entry) hyperviscosity syndrome including but not limited to:

Waldenstrom's macroglobulinemia

Multiple myeloma

Total white blood cell count greater than 80,000/mm(3)

Hematocrit greater than 55%

Platelet count greater than 700,000/mm(3)

Meets criteria of Class III or IV of the New York Heart Association Classification for congestive heart failure patients

Serum creatinine greater than 2.5 mg/dL or requires dialysis

Alternate explanation (as determined by the investigator) for clinical findings (such as structural brain lesion, cerebrovascular accident, or other infectious disease, including confirmed infections with other flaviviruses)

Pregnant or breastfeeding (negative serum or urine pregnancy test within previous 72 hours if woman is not postmenopausal or has not been surgically sterilized)

Investigator's opinion that patient would be unable to adhere to protocol requirements

Receipt of ribavirin, interferon alpha, intravenous immunoglobulin or any investigational drug for treatment of WNV or hepatitis within 15 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2003-09-22; Primary Completion 2007-06-27 (Actual); Study Completion 2007-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] van Swieten JC, Koudstaal PJ, Visser MC, Schouten HJ, van Gijn J. Interobserver agreement for the assessment of handicap in stroke patients. Stroke. 1988 May;19(5):604-7. doi: 10.1161/01.str.19.5.604. PMID 3363593
- [Background] Jennett B, Bond M. Assessment of outcome after severe brain damage. Lancet. 1975 Mar 1;1(7905):480-4. doi: 10.1016/s0140-6736(75)92830-5. PMID 46957
- [Background] McDowell I, Kristjansson B, Hill GB, Hebert R. Community screening for dementia: the Mini Mental State Exam (MMSE) and Modified Mini-Mental State Exam (3MS) compared. J Clin Epidemiol. 1997 Apr;50(4):377-83. doi: 10.1016/s0895-4356(97)00060-7. PMID 9179095
- [Derived] Hart J Jr, Tillman G, Kraut MA, Chiang HS, Strain JF, Li Y, Agrawal AG, Jester P, Gnann JW Jr, Whitley RJ; NIAID Collaborative Antiviral Study Group West Nile Virus 210 Protocol Team. West Nile virus neuroinvasive disease: neurological manifestations and prospective longitudinal outcomes. BMC Infect Dis. 2014 May 9;14:248. doi: 10.1186/1471-2334-14-248. PMID 24884681